CLINICAL TRIAL: NCT03020797
Title: A Clinical Trial to Evaluate the Safety and Efficacy of Fycompa in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1) Enrolment below study target and 2) too many subjects had early termination due to disease progression.
Sponsor: Stony Brook University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Nurcan Gursoy, Clinical Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eisai-01
Record Dates: First submitted 2016-12-15; First posted 2017-01-13 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- perampanel (Experimental): perampanel 2mg QD for 2 weeks perampanel 4mg QD for 2 weeks perampanel 6mg QD for 2 weeks perampanel 8mg QD for 30 weeks
  Interventions: Drug: Perampanel
- placebo (Placebo Comparator): placebo 1 tablet QD for 2 weeks placebo 2 tablets QD for 2 weeks placebo 3 tablets QD for 2 weeks placebo 4 tablets QD for 2 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Perampanel
  Other Names: Fycompa
  Arms: perampanel
Drug: Placebo Oral Tablet
  Arms: placebo

SUMMARY:
This is a pilot trial to test perampanel (Fycompa; Eisai, Inc.) in ALS patients. The investigators will focus on safety and preliminary signs of efficacy. Perampanel is approved by the FDA for treatment of seizures in patients with epilepsy. In this study, perampanel will be used off-label for adults with ALS at an oral medication dose on the low end of the recommended dose range for epilepsy. This study will consist of two treatments arms: perampanel and matching placebo randomized at a 1:1 ratio. Subjects will receive medication for 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of ALS
2. first clinical weakness within past 3 years
3. slow vital capacity >= 60% of predicted within 1 month of treatment
4. may be on stable dose of riluzole for at least 30 days, or otherwise agree to not initiate riluzole for duration of the trial
5. may be on stable dose of edaravone for at least 30 days, otherwise agree to not initiate edaravone for duration of the trial
6. can travel to Stony Brook to receive medical care
7. must have a monitor who can be contacted at regular intervals to report on subject's clinical/psychiatric status

Exclusion Criteria:

1. use of tracheostomy or mechanical ventilation within last 3 months
2. hepatic insufficiency or abnormal liver function
3. renal insufficiency
4. clinically significant psychiatric disorder
5. active malignancy
6. history of HIV, clinically significant chronic hepatitis, or other active infection
7. history of stomach or intestinal surgery or condition that could interfere with absorption, distribution, metabolism or secretion of study drug
8. history of alcohol or substance abuse within 3 months prior to entry (subjects will be instructed to refrain from alcohol during the study)
9. use of strong cytochrome P4503A inhibitors or inducers, anticonvulsants or other drugs known to interact strongly with perampanel.
10. pregnancy or lactation
11. clinically significant medical condition (other than ALS) that would pose a risk to the subject if they were to participate
12. know hypersensitivity to perampanel
13. currently participating, or has participated in a study with an investigation or marketed compound within 3 months of entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 9 months

SECONDARY OUTCOMES:
Efficacy as measured by change in ALSFRS-R score (ALS functional rating scale-revised); | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Gursoy, MD, Principal Investigator — Stony Brook Medicine Dept. of Neurology
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No